CLINICAL TRIAL: NCT04044118
Title: Calorie Restriction Intervention Induces Enterotype-associated BMI Loss in Nonobese Individuals
Acronym: CRDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BGI-Shenzhen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BGI-20170204
Record Dates: First submitted 2019-07-24; First posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-07

CONDITIONS: Healthy Volunteer
Keywords: gut microbiota; calorie restrition dietary intervention
MeSH Terms: interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Caloric Restriction (Experimental): 3-week low calorie diet
  Interventions: Behavioral: Low Calorie Diet

INTERVENTIONS:
Behavioral: Low Calorie Diet — Low Calorie Diet consisted of ~50% calories of a normal-calorie diet (female, 1000kcal/day; male, 1200kcal/day)

SUMMARY:
Calorie restriction (CR), which has the potential effect on weight loss and blood amino acids, has been demonstrated to associate with gut microbiota in humans, especially in obese individuals. However, studies for simultaneously evaluating enterotype-dependent impacts of CR on the gut microbiota and blood amino acids in nonobese individuals are still limited.

Here, 41 nonobese individuals received a 3-week CR diet with approximately 50% fewer calories than a normal diet. The investigators measured individuals' BMI and blood amino acid concentration, along with the gut microbiota before and after the intervention. In this trial, 28 Enterotype Bacteroides (ETB) subjects and 13 Enterotype Prevotella (ETP) subjects were identified before the intervention.

The purpose of this intervention study is to evaluate the effect of calorie restriction on BMI loss, amino acid, and gut microbiota in healthy volunteers of two different enterotypes and provide useful insights for potential application of gut microbiome stratification in personalized nutrition intervention.

DETAILED DESCRIPTION:
1. Volunteer Recruitment

   Volunteer-wanted posters were propagated at the China National Gene Bank in Shenzhen from March to April 2017. A non-obese healthy volunteer was considered if his/her BMI less than 28 kg/m2. 50 individuals met all the criteria and were recruited in this study, and 41 individuals (24 females and 17 males aged 30 ± 6 years old) completed the whole intervention. The study was approved by the institutional review board on bioethics and biosafety of BGI-Shenzhen, Shenzhen (NO. BGI-IRB 17020). All participates were fully informed of the design and purpose of this intervention study and signed a written informed consent letter.
2. Experiment Process

   The study included a one-week run-in period (baseline) and a three-week CR dietary intervention period. During the first week (run-in period), all healthy volunteers consumed their usual diet and were encouraged to avoid yogurt, high-fat foods, and alcohol. The CR diet was comprised of ~50% calories of a normal-calorie diet (female, 1000kcal/day; male, 1200kcal/day). It was designed with carbohydrate, fat, and protein as approximately 55%, 30% and 15% of the total energy intake respectively, according to the Dietary Guidelines for Chinese Residents (2016) and nutritionally balanced and a recent large nutritional study in China. Common foods in low-calorie diets such as rice, vegetables, eggs, pork, and beef were prepared in the investigators' study center to control experimental variables introduced by different foods and calorie estimation errors.

   Traditional Chinese cooking style - boiled, stir-fried and stewed, were applied for the foods. For each meal, digital scales were used to measure the nutritional and caloric values of different foods and total meal for males and females respectively.
3. Sample and Data Collection

BMI, blood and fecal samples of each volunteer were collected at the investigators' study center at baseline and after the 3-week CR intervention. BMI was measured via the clinic scale. The concentrations of 31 amino acids and derivatives in the fasting serum samples were measured by LC-MS/MS. The gut microbial composition was determined using shotgun metagenomics sequencing of fecal DNA.

ELIGIBILITY:
Inclusion Criteria:

* BMI less than 28 kg/m2 and more than 18 kg/m2;
* without antibiotics in the recent 2 months;
* regular eating and lifestyle patterns;
* no international travel in the recent 3 month;
* without hypertension, diabetes mellitus, gastrointestinal disease and other severe auto-immune disease;
* without prebiotic or probiotic supplements in the recent 2 months;

Exclusion Criteria:

* with antibiotics in the recent 2 months;
* Failure to comply with experimental requirement;

Ages: 22 Years to 53 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2018-02-04 (Actual)

PRIMARY OUTCOMES:
change in BMI of all volunteers (n=41) following calorie restriction dietary intervention | at baseline and after 3-week calorie restriction dietary intervention
  BMI was be measured via clinic scale.
different changes in BMI between enterotype Bacteroides (n=28) and enterotype Prevotella (n=13) follow calorie restriction dietary intervention | at baseline and after 3-week calorie restriction dietary intervention
  BMI was be measured via clinic scale.

SECONDARY OUTCOMES:
change in concentration of amino acids of 36 volunteers following calorie restriction dietary intervention | at baseline and after 3-week calorie restriction dietary intervention
  Fasting blood sample for measurement of 31 amino acids
different changes in concentration of 31 amino acids (fasting status) between enterotype Bacteroides (n=25) and enterotype Prevotella (n=11) follow calorie restriction dietary intervention | at baseline and after 3-week calorie restriction dietary intervention
  Fasting blood sample for measurement of 31 amino acids
change in gut microbiota of all volunteers (n=41) following calorie restriction intervention | at baseline and after 3-week calorie restriction dietary intervention
  faecal bacterial composition determined from microbiological cultures and deep metagenomic next-generation sequencing of bacterial DNA in fece
different changes in gut microbiota between enterotype Bacteroides (n=28) and enterotype Prevotella (n=13) follow calorie restriction dietary intervention | at baseline and after 3-week calorie restriction dietary intervention
  faecal bacterial composition determined from microbiological cultures and deep metagenomic next-generation sequencing of bacterial DNA in fece

CONTACTS AND LOCATIONS:
Locations (1):
- BGI-Shenzhen, Guangdong, China, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Statistical analysis plan and analytic code will release
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: analytic code will be available for all the time
Access Criteria: analytic code will be available at github
URL: https://github.com/HuaZou/NonobeseBP

REFERENCES:
- [Background] Wang SS, Lay S, Yu HN, Shen SR. Dietary Guidelines for Chinese Residents (2016): comments and comparisons. J Zhejiang Univ Sci B. 2016 Sep;17(9):649-56. doi: 10.1631/jzus.B1600341. PMID 27604857
- [Background] Redman LM, Huffman KM, Landerman LR, Pieper CF, Bain JR, Muehlbauer MJ, Stevens RD, Wenner BR, Kraus VB, Newgard CB, Kraus WE, Ravussin E. Effect of caloric restriction with and without exercise on metabolic intermediates in nonobese men and women. J Clin Endocrinol Metab. 2011 Feb;96(2):E312-21. doi: 10.1210/jc.2010-1971. Epub 2010 Dec 1. PMID 21123443
- [Background] Santacruz A, Marcos A, Warnberg J, Marti A, Martin-Matillas M, Campoy C, Moreno LA, Veiga O, Redondo-Figuero C, Garagorri JM, Azcona C, Delgado M, Garcia-Fuentes M, Collado MC, Sanz Y; EVASYON Study Group. Interplay between weight loss and gut microbiota composition in overweight adolescents. Obesity (Silver Spring). 2009 Oct;17(10):1906-15. doi: 10.1038/oby.2009.112. Epub 2009 Apr 23. PMID 19390523
- [Background] Ott B, Skurk T, Hastreiter L, Lagkouvardos I, Fischer S, Buttner J, Kellerer T, Clavel T, Rychlik M, Haller D, Hauner H. Effect of caloric restriction on gut permeability, inflammation markers, and fecal microbiota in obese women. Sci Rep. 2017 Sep 20;7(1):11955. doi: 10.1038/s41598-017-12109-9. PMID 28931850
- [Background] Wu GD, Chen J, Hoffmann C, Bittinger K, Chen YY, Keilbaugh SA, Bewtra M, Knights D, Walters WA, Knight R, Sinha R, Gilroy E, Gupta K, Baldassano R, Nessel L, Li H, Bushman FD, Lewis JD. Linking long-term dietary patterns with gut microbial enterotypes. Science. 2011 Oct 7;334(6052):105-8. doi: 10.1126/science.1208344. Epub 2011 Sep 1. PMID 21885731

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/18/NCT04044118/SAP_000.pdf
  • Study Protocol (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/18/NCT04044118/Prot_001.pdf